CLINICAL TRIAL: NCT02757430
Title: EnSite Precision™ Cardiac Mapping System and EnSite Precision™ Software v2.0 Observational Registry
Brief Title: EnSite Precision™ 2.0 Registry
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CIP-10111
Record Dates: First submitted 2016-04-08; First posted 2016-05-02 (Estimated); Results first posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-02

CONDITIONS: Cardiac Arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Cardiac Ablation

SUMMARY:
The objective of this registry is to assess and characterize the use and performance of the EnSite Precision™ Cardiac Mapping System and the EnSite Precision™ Software V2.0 in a variety of electrophysiological (EP) procedures and clinical settings. This registry will assess the clinical performance of the system in a controlled, real-world environment after commercial release.

Up to 500 subjects will be enrolled in up to 50 sites worldwide.

Data will be collected at enrollment/baseline, procedure and pre-discharge. There is no long-term follow-up required for this registry.

The anticipated registry enrollment is about 6-7 months.

DETAILED DESCRIPTION:
The use of the EnSite Precision™ Cardiac Mapping System will be assessed by collecting feedback from physicians/operators through specific questions.

The performance of the EnSite Precision™ Cardiac Mapping System will be assessed by collecting procedure data and adverse events.

A detailed Data Management Plan will be established to ensure consistency of the data. This document will include procedures used for data review, database cleaning, and issuing and resolving data queries. If appropriate, the Data Management Plan may be updated throughout the registry duration. All revisions will be tracked and document controlled.

Case Report Form data will be captured in a validated electronic database management system hosted by St. Jude Medical.

Centralized monitoring will occur through routine internal data review. This monitoring is designed to identify missing and inconsistent data, data outliers, and potential protocol deviations that may be indicative of site non-compliance. On-site monitoring may occur at the discretion of the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for a cardiac EP study and ablation procedure using a 3D mapping system
* Over 18 years of age
* Ability to provide informed consent for registry participation and be willing and able to comply with the protocol described evaluations

Exclusion Criteria:

* Contraindication to anticoagulation
* Presence of thrombus
* Implanted with mechanical prosthetic heart valve
* Recent (<3 months) myocardial Infarction or unstable angina or coronary artery by-pass
* Pregnant or nursing
* Individuals whose willingness to volunteer in a registry, in the judgment of investigator or public authorities, could be unduly influenced by lack of or loss of the autonomy due to immaturity, or mental disability, or adverse personal circumstances, or hierarchical influence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient undergoing a cardiac EP mapping and ablation procedure, using the EnSite™ Precision Cardiac Mapping system, is considered eligible.
Sampling Method: Non-Probability Sample
Enrollment: 515 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Cardinal Massaia di Asti, Asti, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Any patient indicated to undergo a cardiac electrophysiology (EP) mapping and ablation procedure that used the EnSite Precision™ Cardiac Mapping System was considered eligible.
Groups:
- Subjects With EnSite Precision™ Cardiac Mapping: Any patient indicated to undergo a cardiac EP mapping and ablation procedure that used the EnSite Precision™ Cardiac Mapping System was considered eligible. Subjects meeting all inclusion criteria and not meeting any exclusion criteria were enrolled in the study.
Period: Overall Study
Arm/Group | Subjects With EnSite Precision™ Cardiac Mapping
Started | 515
Baseline Visits | 503
EP Mapping/Ablation Procedure | 503
Completed | 503 (Subjects with pre-discharge visit were considered completed.)
Not Completed | 12
Not completed — Physician Decision | 6
Not completed — Inclusion/Exclusion criteria not met | 3
Not completed — No informed consent | 1
Not completed — No procedure performed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Subjects With EnSite Precision™ Cardiac Mapping
Number analyzed (Participants) | 503
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 179
  Male | 324
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 172
  Austria | 23
  Belgium | 2
  Finland | 13
  France | 159
  Germany | 63
  Netherlands | 69
  United Kingdom | 2
Ejection Fraction [Count of Participants; unit: Participants] — 'Abnormal' and 'Normal' ejection fraction defined by physician/Standard Practice
  Participants
    Abnormal per physician/standard of care | 285
    Normal per physician/standard of care | 96
    Not Evaluated | 121
    Not Available | 1
Ejection Fraction [Mean (Standard Deviation); unit: %] — Population: Ejection Fraction provided when evaluated and considered by physician to be abnormal.
  %
    number analyzed (Participants) | 285
    (all) | 54.2 (12.0)
NYHA Heart Failure Classification [Count of Participants; unit: Participants] — New York Heart Association (NYHA) functional classifications are used to classify severity of patient heart failure by placing patients in one of four categories based on how much they are limited during physical activity. Class I is no limitation of physical activity. Class IV is unable to carry on any physical activity without discomfort.
  Participants
    Class I | 108
    Class II | 59
    Class III | 16
    Class IV | 1
    Not Evaluated | 317
    Not Available | 2
Left Atrial Diameter [Mean (Standard Deviation); unit: mm] — Population: Left Atrial Diameter provided when evaluated and considered by physician to be abnormal
  mm
    number analyzed (Participants) | 113
    (all) | 43.1 (8.3)
Left Atrial Volume [Mean (Standard Deviation); unit: ml] — Population: Left Atrial Volume provided when evaluated and considered by physician to be abnormal
  ml
    number analyzed (Participants) | 136
    (all) | 82.3 (42.7)
Indication for Procedure [Count of Participants; unit: Participants]
  Atrial Fibrillation | 277
  Atrial Flutter | 67
  Supraventricular Tachycardia | 96
  Ventricular Tachycardia | 56
  Other | 46

OUTCOME MEASURES:

1. Primary Outcome: Assessment of the EnSite Precision™ Software V2.0 in Terms of Geometry Accuracy
Description: summarizing the count and percentage of patients with accurate geometry
Time Frame: during procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects With EnSite Precision™ Cardiac Mapping
Number analyzed (Participants) | 503
Participants
  Geometry found was anatomically accurate | 461
  Geometry found was not anatomically accurate | 34
  Geometry anatomical accuracy not available | 8

2. Primary Outcome: Mapping Time Associated With (re-)Mapping One or Multiple Arrhythmias in a Single Subject With a Variety of Catheters
Description: mapping time will be summarized (using mean and standard deviation across arrhythmia types, and for each type of arrhythmia as appropriate) for the following modules: Manual AutoMap™ TurboMap™
Time Frame: during procedure
Population: 603 total maps were created in 421 subjects.
Measure: Mean (Standard Deviation); unit: min
Units Other Than Participants: maps
Groups:
- All Maps: All maps created in patients enrolled in the study and who underwent a cardiac EP mapping and ablation procedure that used the EnSite Precision™ Cardiac Mapping System.
Arm/Group | All Maps
Number analyzed (Participants) | 421
Number analyzed (maps) | 603
min
  Manual Map: number analyzed (Participants) | 50
  Manual Map: number analyzed (maps) | 62
  Manual Map | 14.2 (13.9)
  AutoMap: number analyzed (Participants) | 399
  AutoMap: number analyzed (maps) | 526
  AutoMap | 13.1 (11.9)
  TurboMap: number analyzed (Participants) | 12
  TurboMap: number analyzed (maps) | 13
  TurboMap | 6.6 (5.7)
  Other: number analyzed (Participants) | 2
  Other: number analyzed (maps) | 2
  Other | 4.0 (1.4)

3. Primary Outcome: Mapping Time Associated With (re-)Mapping One or Multiple Arrhythmias in a Single Subject With a Variety of Catheters With Manual Mapping
Description: mapping time will be summarized (using mean and standard deviation across arrhythmia types, and for each type of arrhythmia as appropriate) for the following modules: Manual
Time Frame: during procedure
Population: 62 total Manual maps were created.
Measure: Mean (Standard Deviation); unit: min
Units Other Than Participants: manual maps
Groups:
- All Manual Maps: All manual maps created in patients enrolled in the study and who underwent a cardiac EP mapping and ablation procedure that used the EnSite Precision™ Cardiac Mapping System.
Arm/Group | All Manual Maps
Number analyzed (Participants) | 50
Number analyzed (manual maps) | 62
min
  Sinus Rhythm: number analyzed (Participants) | 6
  Sinus Rhythm: number analyzed (manual maps) | 7
  Sinus Rhythm | 11.5 (9.8)
  Atrial Fibrillation: number analyzed (Participants) | 1
  Atrial Fibrillation: number analyzed (manual maps) | 1
  Atrial Fibrillation | 20.0 (NA) — No standard deviation for N of 1
  Atrial Flutter: number analyzed (Participants) | 5
  Atrial Flutter: number analyzed (manual maps) | 6
  Atrial Flutter | 8.8 (4.3)
  Atrial Tachycardia: number analyzed (Participants) | 12
  Atrial Tachycardia: number analyzed (manual maps) | 14
  Atrial Tachycardia | 18.3 (18.2)
  Atrioventricular Reentry Tachycardia: number analyzed (Participants) | 2
  Atrioventricular Reentry Tachycardia: number analyzed (manual maps) | 2
  Atrioventricular Reentry Tachycardia | 10.0 (0.0)
  Atrioventricular Nodal Reentry Tachycardia: number analyzed (Participants) | 6
  Atrioventricular Nodal Reentry Tachycardia: number analyzed (manual maps) | 8
  Atrioventricular Nodal Reentry Tachycardia | 3.6 (3.3)
  Ventricular Tachycardia: number analyzed (Participants) | 6
  Ventricular Tachycardia: number analyzed (manual maps) | 8
  Ventricular Tachycardia | 23.4 (19.3)
  Other: number analyzed (Participants) | 14
  Other: number analyzed (manual maps) | 16
  Other | 14.6 (11.6)

4. Primary Outcome: Mapping Time Associated With (re-)Mapping One or Multiple Arrhythmias in a Single Subject With a Variety of Catheters With AutoMap Module Mapping
Description: mapping time will be summarized (using mean and standard deviation across arrhythmia types, and for each type of arrhythmia as appropriate) for the following modules: AutoMap module
Time Frame: during procedure
Population: 526 total AutoMap Module maps were created.
Measure: Mean (Standard Deviation); unit: min
Units Other Than Participants: AutoMap Module Maps
Groups:
- All AutoMap Module Maps: All AutoMap module maps created in patients enrolled in the study and who underwent a cardiac EP mapping and ablation procedure that used the EnSite Precision™ Cardiac Mapping System.
Arm/Group | All AutoMap Module Maps
Number analyzed (Participants) | 399
Number analyzed (AutoMap Module Maps) | 526
min
  Sinus Rhythm: number analyzed (Participants) | 264
  Sinus Rhythm: number analyzed (AutoMap Module Maps) | 297
  Sinus Rhythm | 14.3 (13.5)
  Atrial Fibrillation: number analyzed (Participants) | 51
  Atrial Fibrillation: number analyzed (AutoMap Module Maps) | 58
  Atrial Fibrillation | 11.3 (5.4)
  Atrial Flutter: number analyzed (Participants) | 48
  Atrial Flutter: number analyzed (AutoMap Module Maps) | 59
  Atrial Flutter | 10.1 (7.3)
  Atrial Tachycardia: number analyzed (Participants) | 27
  Atrial Tachycardia: number analyzed (AutoMap Module Maps) | 42
  Atrial Tachycardia | 8.4 (5.8)
  Atrioventricular Reentry Tachycardia: number analyzed (Participants) | 1
  Atrioventricular Reentry Tachycardia: number analyzed (AutoMap Module Maps) | 1
  Atrioventricular Reentry Tachycardia | 6.0 (NA) — No standard deviation for N of 1
  Atrioventricular Nodal Reentry Tachycardia: number analyzed (Participants) | 2
  Atrioventricular Nodal Reentry Tachycardia: number analyzed (AutoMap Module Maps) | 2
  Atrioventricular Nodal Reentry Tachycardia | 11.0 (1.4)
  Ventricular Tachycardia: number analyzed (Participants) | 22
  Ventricular Tachycardia: number analyzed (AutoMap Module Maps) | 26
  Ventricular Tachycardia | 16.3 (16.2)
  Other: number analyzed (Participants) | 37
  Other: number analyzed (AutoMap Module Maps) | 41
  Other | 14.3 (10.8)

5. Primary Outcome: Mapping Time Associated With (re-)Mapping One or Multiple Arrhythmias in a Single Subject With a Variety of Catheters With TurboMap Module Mapping
Description: mapping time will be summarized (using mean and standard deviation across arrhythmia types, and for each type of arrhythmia as appropriate) for the following modules: TurboMap module
Time Frame: during procedure
Population: 13 total TurboMap Module maps were created.
Measure: Mean (Standard Deviation); unit: min
Units Other Than Participants: TurboMap Module Maps
Groups:
- All TurboMap Module Maps: All TurboMap module maps created in patients enrolled in the study and who underwent a cardiac EP mapping and ablation procedure that used the EnSite Precision™ Cardiac Mapping System.
Arm/Group | All TurboMap Module Maps
Number analyzed (Participants) | 12
Number analyzed (TurboMap Module Maps) | 13
min
  Sinus Rhythm: number analyzed (Participants) | 3
  Sinus Rhythm: number analyzed (TurboMap Module Maps) | 3
  Sinus Rhythm | 4.3 (1.2)
  Atrial Fibrillation: number analyzed (Participants) | 1
  Atrial Fibrillation: number analyzed (TurboMap Module Maps) | 1
  Atrial Fibrillation | 17.0 (NA) — no standard deviation for N of 1
  Atrial Flutter: number analyzed (Participants) | 4
  Atrial Flutter: number analyzed (TurboMap Module Maps) | 4
  Atrial Flutter | 3.3 (0.5)
  Atrial Tachycardia: number analyzed (Participants) | 2
  Atrial Tachycardia: number analyzed (TurboMap Module Maps) | 2
  Atrial Tachycardia | 8.0 (9.9)
  Other: number analyzed (Participants) | 2
  Other: number analyzed (TurboMap Module Maps) | 3
  Other | 9.0 (7.2)

6. Primary Outcome: Point Density Associated With (re-)Mapping One or Multiple Arrhythmias in a Single Subject With a Variety of Catheters
Description: mapping points collected and used will be summarized (using mean and standard deviation across arrhythmia types, and for each type of arrhythmia as appropriate)
Time Frame: during procedure
Population: 606 total maps with mapping points collected available were created in 421 subjects.
Measure: Mean (Standard Deviation); unit: mapping points collected
Units Other Than Participants: maps
Groups:
- All Maps With Mapping Points Collected: All maps with number of mapping points collected available created in patients enrolled in the study and who underwent a cardiac EP mapping and ablation procedure that used the EnSite Precision™ Cardiac Mapping System.
Arm/Group | All Maps With Mapping Points Collected
Number analyzed (Participants) | 421
Number analyzed (maps) | 606
mapping points collected
  All Arrhythmias | 2074.7 (3377.2)
  Sinus Rhythm: number analyzed (Participants) | 269
  Sinus Rhythm: number analyzed (maps) | 308
  Sinus Rhythm | 2396.0 (3638.5)
  Atrial Fibrillation: number analyzed (Participants) | 52
  Atrial Fibrillation: number analyzed (maps) | 60
  Atrial Fibrillation | 3124.3 (3253.4)
  Atrial Flutter: number analyzed (Participants) | 53
  Atrial Flutter: number analyzed (maps) | 70
  Atrial Flutter | 2484.3 (4440.9)
  Atrial Tachycardia: number analyzed (Participants) | 35
  Atrial Tachycardia: number analyzed (maps) | 58
  Atrial Tachycardia | 1957.0 (2331.0)
  Atrioventricular Reentry Tachycardia: number analyzed (Participants) | 2
  Atrioventricular Reentry Tachycardia: number analyzed (maps) | 2
  Atrioventricular Reentry Tachycardia | 143.5 (169.0)
  Arioventricular Nodal Reentry Tachycardia: number analyzed (Participants) | 8
  Arioventricular Nodal Reentry Tachycardia: number analyzed (maps) | 10
  Arioventricular Nodal Reentry Tachycardia | 95.0 (237.6)
  Ventricular Tachycardia: number analyzed (Participants) | 25
  Ventricular Tachycardia: number analyzed (maps) | 36
  Ventricular Tachycardia | 841.9 (1698.7)
  Other: number analyzed (Participants) | 49
  Other: number analyzed (maps) | 62
  Other | 208.4 (438.0)

7. Primary Outcome: Point Density Associated With (re-)Mapping One or Multiple Arrhythmias in a Single Subject With a Variety of Catheters
Description: as for outcome 6
Time Frame: during procedure
Population: 606 total maps with mapping points used available were created in 421 subjects.
Measure: Mean (Standard Deviation); unit: mapping points used
Units Other Than Participants: maps
Groups:
- All Maps With Mapping Points Used: All maps with number of mapping points used available created in patients enrolled in the study and who underwent a cardiac EP mapping and ablation procedure that used the EnSite Precision™ Cardiac Mapping System.
Arm/Group | All Maps With Mapping Points Used
Number analyzed (Participants) | 421
Number analyzed (maps) | 606
mapping points used
  All Arrhythmias | 781.9 (1062.1)
  Sinus Rhythm: number analyzed (Participants) | 269
  Sinus Rhythm: number analyzed (maps) | 308
  Sinus Rhythm | 954.5 (1245.6)
  Atrial Fibrillation: number analyzed (Participants) | 52
  Atrial Fibrillation: number analyzed (maps) | 60
  Atrial Fibrillation | 1127.3 (801.6)
  Atrial Flutter: number analyzed (Participants) | 53
  Atrial Flutter: number analyzed (maps) | 70
  Atrial Flutter | 828.8 (983.4)
  Atrial Tachycardia: number analyzed (Participants) | 35
  Atrial Tachycardia: number analyzed (maps) | 58
  Atrial Tachycardia | 612.3 (663.6)
  Atrioventricular Reentry Tachycardia: number analyzed (Participants) | 2
  Atrioventricular Reentry Tachycardia: number analyzed (maps) | 2
  Atrioventricular Reentry Tachycardia | 85.5 (103.9)
  Arioventricular Nodal Reentry Tachycardia: number analyzed (Participants) | 8
  Arioventricular Nodal Reentry Tachycardia: number analyzed (maps) | 10
  Arioventricular Nodal Reentry Tachycardia | 56.7 (134.2)
  Ventricular Tachycardia: number analyzed (Participants) | 25
  Ventricular Tachycardia: number analyzed (maps) | 36
  Ventricular Tachycardia | 318.1 (623.7)
  Other: number analyzed (Participants) | 49
  Other: number analyzed (maps) | 62
  Other | 104.3 (182.6)

8. Primary Outcome: Assessment of the EnSite Precision™ Software V2.0 in Terms of System Stability
Description: summarizing the count and percentage of patients with overall system stability
Time Frame: during procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects With EnSite Precision™ Cardiac Mapping
Number analyzed (Participants) | 503
Participants
  System was stable throughout the procedure | 455
  System was not stable throughout the procedure | 46
  Stability throughout the procedure not available | 2

9. Primary Outcome: Assessment of the EnSite Precision™ Software V2.0 in Terms of Unrecoverable Shifts
Description: summarizing the count and percentage of patients with unrecoverable shifts
Time Frame: during procedure
Population: 46 procedures with system not stable throughout the procedure
Measure: Count of Participants; unit: Participants
Groups:
- Procedures With Unstable Maps: System stability throughout the procedure was assessed. System was not stable throughout the procedure in 46 procedures.
Arm/Group | Procedures With Unstable Maps
Number analyzed (Participants) | 46
Participants
  Map could be recovered | 36
  Map could not be recovered | 10

10. Secondary Outcome: EnSite Precision™ Cardiac Mapping System Assessment
Description: Count and percentage of subjects in whom the mapping system was reported to be excellent, very good, good, poor and N/A
Time Frame: during procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects With EnSite Precision™ Cardiac Mapping
Number analyzed (Participants) | 503
Participants
  Excellent | 153
  Very Good | 202
  Good | 139
  Poor | 8
  Not Applicable | 1

11. Secondary Outcome: EnSite Precision™ Cardiac Mapping System Assessment
Description: Overall procedure time summarized using mean and standard deviation
Time Frame: during procedure
Population: 501 subjects had procedure time available
Measure: Mean (Standard Deviation); unit: mins
Arm/Group | Subjects With EnSite Precision™ Cardiac Mapping
Number analyzed (Participants) | 501
mins | 116.8 (52.2)

12. Secondary Outcome: Clinical Utility and Ease of Use of the Automated Radiofrequency Marker Placement
Description: Count and percentage of subjects where the AutoMark feature assisted in identifying gaps in lesion lines
Time Frame: during procedure
Population: 117 subjects had gaps identified in the lesion line
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects With Identified Gaps in Lesion Line: All subjects with ablation procedure performed and gap identified in lesion line.
Arm/Group | All Subjects With Identified Gaps in Lesion Line
Number analyzed (Participants) | 117
Participants
  AutoMark assisted in identifying gaps | 34
  AutoMark did not assist in identifying gaps | 83

13. Secondary Outcome: Clinical Utility and Ease of Use of the Automated Radiofrequency Marker Placement
Description: Count and percentage of subjects where the AutoMark feature was easy to use
Time Frame: during procedure
Population: 373 procedures used AutoMark
Measure: Count of Participants; unit: Participants
Groups:
- Procedures With AutoMark Feature Used: All procedures in which the EnSite(TM) AutoMark feature was used
Arm/Group | Procedures With AutoMark Feature Used
Number analyzed (Participants) | 373
Participants
  AutoMark feature was easy to use | 352
  AutoMark feature was not easy to use | 4
  AutoMark Feature ease of use not available | 17

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the beginning of the procedure through the Pre-discharge visit (maximum of 7 days after procedure).
Description: Any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device under study.
  This definition includes events related to the investigational medical device or the comparator.
  This definition includes events related to the procedures involved.
Arm/Group | Subjects With EnSite Precision™ Cardiac Mapping
All-Cause Mortality (participants affected / at risk) | 0/503
Serious Adverse Events (participants affected / at risk) | 10/503
Other Adverse Events (participants affected / at risk) | 2/503
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With EnSite Precision™ Cardiac Mapping (N=503)
Non-Sustained Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Recurrence of Atrial Fibrillation (Cardiac disorders) | 1 (1)
Recurrent Arrhythmia (Cardiac disorders) | 1 (1)
Esophageal Lesion (Gastrointestinal disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachy-Brady Syndrome (Cardiac disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Tamponade (Cardiac disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With EnSite Precision™ Cardiac Mapping (N=503)
Atrioventricular Nodal Reentrant Tachycardia (Cardiac disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/30/NCT02757430/Prot_SAP_ICF_000.pdf